CLINICAL TRIAL: NCT00679081
Title: A Prospective, Randomized, Controlled Pilot Study of CelTx(TM) (Apligraf®) as an Alternative to Tissue From the Palate in the Treatment of Gingival Recession Requiring Root Coverage
Brief Title: A Pilot Study of CelTx(TM) (Apligraf®) in the Treatment of Gingival Recession Requiring Root Coverage
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-PER-004-CTX
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2011-11-21 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CelTx (Experimental): CelTx
  Interventions: Device: CelTx
- Autologous CTG (Active Comparator): Autologous sub-epithelial connective tissue graft
  Interventions: Other: Autologous sub-epithelial connective tissue graft

INTERVENTIONS:
Device: CelTx — Single application; split-mouth design
  Arms: CelTx
Other: Autologous sub-epithelial connective tissue graft — Single application; split-mouth design
  Arms: Autologous CTG

SUMMARY:
The purpose of this study is to evaluate CelTx as an alternative to tissue from the palate in the treatment of subjects with Miller Class I or II recession defects who desire root coverage. It is anticipated that this study will demonstrate that CelTx is a safe alternative to palatal tissue and demonstrate potential to enhance oral soft tissue regeneration and wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age but no more than 70 years of age.
* Subject has at least two non-adjacent teeth in contralateral quadrants of the same jaw with Miller Class I or II buccal recession (≥ 3 mm) that requires soft tissue grafting. (Teeth may be treated with a maximum difference of 2 mm with respect to depth and width).
* Females of childbearing potential must have a documented negative urine pregnancy test and must agree to continue acceptable methods of contraception for 6 months post surgery.
* Subjects must have read, understood and signed an institutional review board (IRB)-approved Informed Consent Form (ICF).
* Subjects must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

* Subject has extremely prominent root surfaces (> 1/2 the diameter of the root facial to cortical plate).
* Subject has interproximal attachment loss beyond the CEJ.
* Subject with teeth that have a Miller Grade 2 or higher mobility.
* Subjects with Class V restorations.
* Subjects with crowns on the teeth selected for treatment.
* Subjects who have had endodontic therapy in the last 6 months on the teeth selected for treatment.
* Subjects who have used any tobacco product within the past 3 months.
* Subjects with only molar teeth suitable for soft tissue grafting.
* Subject has probing pocket depth >/= 4 mm at either surgical site.
* Female subjects who are pregnant or lactating.
* Subjects with any systemic conditions (i.e., uncontrolled diabetes mellitus, cancer, HIV, bone metabolic diseases) that could compromise wound healing and preclude periodontal surgery.
* Subjects who are currently receiving or have received within two months prior to study entry, systemic corticosteroids, immunosuppressive agents, radiation therapy, and/or chemotherapy which could compromise wound healing and preclude periodontal surgery.
* Subjects with the presence of acute infectious lesions.
* Subjects taking intramuscular or intravenous bisphosphonates.
* Subjects with a known hypersensitivity to bovine collagen and/or iodine (shellfish allergy).
* Subjects who have received an investigational drug, device or biological/bioactive treatment within 30 days prior to study enrollment (medical or dental).
* Subjects previously treated with Apligraf/CelTx, Dermagraft or any other cell-based product, including autologous tissue at the target site(s) or immediately adjacent teeth.
* Subjects, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGuire, DDS, Principal Investigator — Perio Health Professionals, PLLC
Locations (1):
- Perio Health Professionals, PLLC, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CelTx and Autologous CTG; Split-mouth Design: Enrolled subjects had 2 non-adjacent teeth in contralateral quadrants of the same jaw identified and randomized to treatment with CelTx or autologous sub-epithelial connective tissue graft (CTG). Either a folded or a single layer of CelTx or autologous sub-epithelial CTG was applied to the teeth selected for treatment according to the randomization scheme; only 1 tooth was treated per quadrant. The harvested autologous sub-epithelial CTG was shaped to fit the recipient site and was similar in size to CelTx. Surgical site preparation and CelTx and autologous sub-epithelial CTG placement were the same for both treatment sites.
Period: Overall Study
Arm/Group | CelTx and Autologous CTG; Split-mouth Design
Started | 15 (Study design was within-subject control.)
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | CelTx and Autologous CTG; Split-mouth Design
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 42.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  Asian | 3
  American Indian or Alaska Native | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of Adverse Events (AEs)
Description: Adverse events were collected at every visit throughout the 6 month duration.
  An AE is defined as any adverse change in the subject's medical status when compared with the subject's baseline condition, whether or not the event is related to the study device or a study procedure; or an exacerbation (either in frequency or severity) in a subject's pre-existing condition.
Time Frame: 6-month
Measure: Number; unit: participants
Groups:
- CelTx Site: Adverse events occurring at the CelTx site
- Graft Site: Adverse events occurring at the autologous sub-epithelial connective tissue graft site
- Other Location: Adverse events occurring at a site other than the CelTx or Autologous graft sites
Arm/Group | CelTx Site | Graft Site | Other Location
Number analyzed (Participants) | 15 | 15 | 15
participants | 2 | 2 | 8

2. Secondary Outcome: Periodontal Health Measures
Time Frame: 6-months
Reporting Status: Not Posted

3. Secondary Outcome: Aesthetic Measures
Time Frame: 6-months
Reporting Status: Not Posted

4. Secondary Outcome: Post-Surgical Subject Comfort Measures
Time Frame: 4-weeks
Reporting Status: Not Posted

5. Secondary Outcome: Subject Preference Measures
Time Frame: 6-months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CelTx Site | Graft Site | Other Location
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 2/15 | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CelTx Site (N=15) | Graft Site (N=15) | Other Location (N=15)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral Mucosa Erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired Healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis Infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Gingival Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Suture Related Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to suboptimal clinical outcomes. Due to two study design changes, the data could not be combined and analyzed for effectiveness (ie, no secondary effectiveness endpoints were tested).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for at least 30 days in advance of public release. The sponsor can request removal of any confidential or proprietary information provided by sponsor and extend such review period for another 90 days to file patent applications or take other steps to protect the sponsor's intellectual property interests.